CLINICAL TRIAL: NCT01808794
Title: Clinical, Radiographic, and Histological Comparison of Healing After Alveolar Ridge Preservation Using Bone Allograft With Two Different Xenogeneic Membranes
Brief Title: Comparison of Two Different Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUSDM10551; 10551 (Other: Tufts University IRB)
Record Dates: First submitted 2013-03-05; First posted 2013-03-11 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Partial Edentulism
Keywords: membranes; Mucograft; Dynamatrixw; ridge; preservation; bone; allograft; extraction; site; healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucograft (Active Comparator): Placement of randomized membrane on half of subjects Mucograft
  Interventions: Device: Mucograft
- Dynamatrix (Active Comparator): Placement of randomized membrane on half of subjects Dynamatrix Membrane Placement
  Interventions: Device: Dynamatrix

INTERVENTIONS:
Device: Mucograft — Mucograft Collagen Matrix
  Other Names: 510(k) #K073711
  Arms: Mucograft
Device: Dynamatrix — Dynamatrix
  Other Names: 510(k) #K082058
  Arms: Dynamatrix

SUMMARY:
The purpose of the study is to compare one material called "Mucograft" with another material called "Dynamatrix." These materials are used as a type of a barrier (made from pig material also known as porcine material) in a preservation technique to increase the thickness and width of tissues at a tooth extraction site. The investigators want to see if one works better than the other or if they work equally as well. These materials are made up of collagens, which are naturally occurring proteins found in the skin, specifically connective tissue. Dynamatrix is made up of many types of collagens whereas Mucograft is only made of fewer collagens. These materials have been given something called a 510(k) status by the FDA. This means that the FDA determines them to be equivalent to another product that they have previously approved. You will be put into one of two groups at random, and will not know which one you are in. Like flipping a coin, you will have a 50/50 chance to be in either one of the two groups. You will either be in a group using Mucograft or in a group using Dynamatrix. Both of these materials are regularly used in the dental clinics.

DETAILED DESCRIPTION:
A) Aim/Hypothesis/Objective The objective of this study is to compare two different membranes, Mucograft and Dynamatrix, clinically, radiographically, and histologically when used for the ridge preservation procedure in combination with bone allograft at the extraction site in terms of soft and hard tissue remodeling after 4 months healing period.

Hypothesis

1. MucograftTM will exhibit greater increase or preservation of the thickness and width of keratinized tissue than DynamatrixTM at the extraction site.
2. MucograftTM will exhibit greater preservation of the alveolar bone width and height than DynamatrixTM at the extraction site.
3. MucograftTM will exhibit greater preservation of the soft and hard tissue height than DynamatrixTM at the adjacent teeth.
4. MucograftTM will exhibit a better outcome than DynamatrixTM in the histological and histomorphometric results of the soft and hard tissue healing.

Specific Aims

1. Primary aim The primary aim is to compare MucograftTM when used as a barrier membrane in the ridge preservation technique to increase or preserve the thickness and width of keratinized tissue at the extraction site in comparison to DynamatrixTM.
2. Secondary aims

The secondary aims are to compare clinically, radiographically, and histologically MucograftTM with DynamatrixTM in relation to:

1. Changes of the alveolar bone height and width at the extraction site.
2. Changes of the soft and hard tissues at the adjacent teeth.
3. Histological and histomorphometric assessment of the soft and hard tissue healing at the extraction site.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Have unsalvageable non-adjacent non-molar teeth: maxillary incisors, canines, and premolars, and mandibular canines and premolars that require an extraction with bone augmentation planned for delayed implant placement. If a subject has multiple teeth to be extracted, only one tooth will be included in the study.
3. Patients who are currently treatment planned in the Tufts University School of Dental Medicine (TUSDM) periodontology clinic to receive bone augmentation and delayed implant placement and meet all medical and dental requirements of the TUSDM periodontology clinic for periodontal surgery (e.g., subjects with no diseases or medication allergies contraindicating periodontal surgery).
4. Display no evidence of acute periodontal infection: e.g., abscess, suppuration, severe swelling and/or spontaneous bleeding.
5. Smoke less than 10 cigarettes per day.
6. Not participating in any other dental research study for the duration of this study.

Exclusion Criteria:

1. Have any known disease that interferes with periodontal surgery and would not allow the patient to be treatment planned for the procedures in the TUSDM periodontology clinic (e.g., severe anemia, low white blood cell count, bleeding or coagulation disorder, uncontrolled hypertension, recent myocardial infarction (within 6 months of enrollment), poorly controlled diabetes, HIV/AIDS (self-reported), history of or currently undergoing head and neck radiation, history of or currently taking bisphosphonates).
2. Have a history of severe psychological conditions or limited mental capacity.
3. Be a pregnant or lactating female (self-reported) (following TUSDM periodontology clinic guidelines elective surgical procedures and radiographs/CBCT scans are usually postponed until after delivery).
4. Individuals opposed to having porcine derived materials placed in their mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hanley, DMD, Principal Investigator — TUSDM; Youngsoo Kim, DDS, Study Director — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available
Period: Overall Study
Arm/Group | Mucograft | Dynamatrix
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mucograft | Dynamatrix | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Compare Barrier Membranes by Examining Keratinized Tissue
Description: The primary aim is to compare MucograftTM when used as a barrier membrane in the ridge preservation technique to increase or preserve the thickness and width of keratinized tissue at the extraction site in comparison to DynamatrixTM.
Time Frame: 4-6 Months after surgical procedure
Population: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available.
Arm/Group | Mucograft | Dynamatrix
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Alveolar Bone Height
Description: Compare clinically, radiographically, and histologically MucograftTM with DynamatrixTM in relation to changes of the alveolar bone height at the extraction site.
Time Frame: 4-6 Months after surgical procedure
Population: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available.
Arm/Group | Mucograft | Dynamatrix
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available.
Description: The Study PI has passed away. All efforts to locate study data have been exhausted and there is no study data available.
Arm/Group | Mucograft | Dynamatrix
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No